CLINICAL TRIAL: NCT05339971
Title: Modified Surgical Technique for Lateral Block Augmentation Prior to Implant Installation - A Pilot Study on 10 Patients With Histological Assessment
Brief Title: Modified Surgical Technique for Lateral Block Augmentation Prior to Implant Installation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Kristina Bertl, Principal Investigator, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1401/2016
Record Dates: First submitted 2022-04-09; First posted 2022-04-21 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Bone Augmentation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- block perforation (Experimental)
  Interventions: Other: block perforation

INTERVENTIONS:
Other: block perforation — The bone block used for lateral bone augmentation will be perforated several times.

SUMMARY:
Evaluation of the surgical result (augmentation volume, proportion of newly formed bone) after perforation of the bone block in the course of lateral block augmentation prior to planned implant installation.

ELIGIBILITY:
Inclusion Criteria:

* single tooth gap in need of lateral bone augmentation prior to implant installation

Exclusion Criteria:

* untreated periodontal disease
* systemic disease and/or medication intake with significant effect on bone healing

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-12-07 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Histomorphometry | at implant installation (approximately 6 months after augmentation)
  % of new bone formation
Radiographic | 6 months after block augmentation
  Volume gain (mm3) after block augmentation at the buccal aspect
Radiographic | 12 months after block augmentation
  Volume gain (mm3) after block augmentation at the buccal aspect